CLINICAL TRIAL: NCT06984237
Title: Psoriasis and Periodontitis Are Chronic Inflammatory Diseases That May Share Common Immunopathogenic Pathways. TNF-α, IL-17A, and YKL-40 Are Inflammatory Biomarkers Associated With Both Conditions. This Study Aims to Evaluate the Levels of These Markers in Saliva and Serum of Individuals With Psoriasis, Considering Their Periodontal Status, to Investigate a Potential Link Between the Two Diseases
Brief Title: Evaluation of Salivary and Serum Levels of TNF-α, IL-17A, and YKL-40 in Individuals With Psoriasis
Status: Active, not recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hazal Durmus, DDS, Akdeniz University
Other Study IDs: AkdenizU Psoriasis
Record Dates: First submitted 2025-05-08; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Psoriasis
Keywords: TNF-α; IL-17A; YKL-40; salivary; serum
MeSH Terms: conditions — Periodontitis; Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1. Group: Healthy (H): 1. Group: Healthy (H):Systemically and periodontally healthy individuals (H)
  Interventions: Diagnostic Test: TNF-α Analysis in saliva; Diagnostic Test: IL-17A analysis in saliva; Diagnostic Test: YKL-40 Analysis in saliva; Diagnostic Test: TNF-α analysis in serum; Diagnostic Test: IL-17A analysis in serum; Diagnostic Test: YKL-40 analysis in serum; Diagnostic Test: Clinical periodontal evaluation
- 2. Group: Control Gingivitis(CG): 2. Group: Control Gingivitis(CG): Systemically healthy individuals with gingivitis
  Interventions: Diagnostic Test: TNF-α Analysis in saliva; Diagnostic Test: IL-17A analysis in saliva; Diagnostic Test: YKL-40 Analysis in saliva; Diagnostic Test: TNF-α analysis in serum; Diagnostic Test: IL-17A analysis in serum; Diagnostic Test: YKL-40 analysis in serum; Diagnostic Test: Clinical periodontal evaluation
- 3. Group: Control Periodontitis(CP): 3. Group: Control Periodontitis(CP): Systemically healthy individuals with periodontitis
  Interventions: Diagnostic Test: TNF-α Analysis in saliva; Diagnostic Test: IL-17A analysis in saliva; Diagnostic Test: YKL-40 Analysis in saliva; Diagnostic Test: TNF-α analysis in serum; Diagnostic Test: IL-17A analysis in serum; Diagnostic Test: YKL-40 analysis in serum; Diagnostic Test: Clinical periodontal evaluation
- 4. Group: Psoriasis Gingivitis(PG): 4. Group: Psoriasis Gingivitis(PG): Individuals with psoriasis and gingivitis
  Interventions: Diagnostic Test: TNF-α Analysis in saliva; Diagnostic Test: IL-17A analysis in saliva; Diagnostic Test: YKL-40 Analysis in saliva; Diagnostic Test: TNF-α analysis in serum; Diagnostic Test: IL-17A analysis in serum; Diagnostic Test: YKL-40 analysis in serum; Diagnostic Test: Clinical periodontal evaluation
- 5. Group: Psoriasis Periodontitis (PP): 5. Group: Psoriasis Periodontitis (PP): Individuals with psoriasis and periodontitis
  Interventions: Diagnostic Test: TNF-α Analysis in saliva; Diagnostic Test: IL-17A analysis in saliva; Diagnostic Test: YKL-40 Analysis in saliva; Diagnostic Test: TNF-α analysis in serum; Diagnostic Test: IL-17A analysis in serum; Diagnostic Test: YKL-40 analysis in serum; Diagnostic Test: Clinical periodontal evaluation

INTERVENTIONS:
Diagnostic Test: TNF-α Analysis in saliva — Unstimulated whole saliva samples will be collected in the morning, at least one day after periodontal examination. Participants will be instructed to refrain from eating, drinking, brushing, or chewing gum for at least one hour before collection. The samples will be centrifuged at 1500 rpm for 10 minutes, and the supernatants will be stored at -80°C until analysis. TNF-α levels will be measured using ELISA.
Diagnostic Test: IL-17A analysis in saliva — Unstimulated whole saliva samples will be collected in the morning, at least one day after periodontal examination. Participants will be asked to avoid eating, drinking, brushing their teeth, or chewing gum for at least one hour prior to sampling. The samples will be centrifuged at 1500 rpm for 10 minutes, and the supernatants will be stored at -80°C until analysis. IL-17A levels will be determined using ELISA.
Diagnostic Test: YKL-40 Analysis in saliva — Unstimulated whole saliva samples will be obtained from participants in the morning, at least one day after the periodontal clinical assessment. They will be instructed not to eat, drink, chew gum, or brush their teeth for at least one hour before collection. Samples will be centrifuged at 1500 rpm for 10 minutes, and the clear supernatants will be stored at -80°C until the time of analysis. YKL-40 levels will be measured using ELISA.
Diagnostic Test: TNF-α analysis in serum — A total of 8 mL of venous blood will be collected from the antecubital fossa of seated participants. Samples will be transferred into BD Vacutainer® SST™ II Advance serum separator tubes containing acrylic gel and will be allowed to clot for 30 minutes at room temperature. The samples will then be centrifuged at 1500 rpm for 10 minutes at 18-25°C. The resulting serum will be transferred into Eppendorf tubes using a Pasteur pipette and will be stored at -80°C until analysis. TNF-α levels will be measured using ELISA.
Diagnostic Test: IL-17A analysis in serum — A total of 8 mL of venous blood will be obtained from the antecubital fossa of participants in a seated position. After collection, the blood will be placed into BD Vacutainer® SST™ II Advance tubes with acrylic gel and will rest for 30 minutes to allow clotting. The samples will be centrifuged at 1500 rpm for 10 minutes at 18-25°C. The serum will be extracted using a Pasteur pipette and stored in Eppendorf tubes at -80°C until analysis. IL-17A levels will be analyzed using ELISA.
Diagnostic Test: YKL-40 analysis in serum — Venous blood (8 mL) will be drawn from the antecubital fossa of seated participants. The samples will be placed in BD Vacutainer® SST™ II Advance tubes containing acrylic gel and will be left to clot for 30 minutes at room temperature. Following this, the samples will be centrifuged at 1500 rpm for 10 minutes at 18-25°C. The supernatant serum will be separated with a Pasteur pipette and transferred into Eppendorf tubes. All samples will be stored at -80°C until analysis. YKL-40 levels will be measured using ELISA.
Diagnostic Test: Clinical periodontal evaluation — Clinical periodontal parameters will be recorded from participants who meet the inclusion criteria. The following indices will be measured from all teeth present in the oral cavity: Plaque Index (PI; Silness & Löe, 1964), Probing Pocket Depth (PPD), Clinical Attachment Level (CAL), and Bleeding on Probing (BOP). Radiographic evaluations will also be performed. All measurements will be conducted by the same calibrated clinician (HD) using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA).

SUMMARY:
Background: Periodontitis is a chronic inflammatory disease triggered by microbial infections that lead to the destruction of tissues supporting the teeth. Psoriasis is a chronic skin condition characterized by excessive proliferation and abnormal differentiation of keratinocytes. Due to the presence of similar inflammatory mechanisms, an immunological relationship between psoriasis and periodontal disease has been hypothesized. To explore this relationship, the levels of TNF-α, IL-17A, and YKL-40 in saliva and serum will be examined in both systemically healthy individuals and individuals with psoriasis.

Methods: The study will include five distinct groups based on systemic and periodontal conditions:

1. systemically and periodontally healthy individuals (H),
2. systemically healthy individuals with gingivitis (Control Gingivitis, CG),
3. systemically healthy individuals with periodontitis (Control Periodontitis, CP),
4. individuals with psoriasis and gingivitis (Psoriasis Gingivitis, PG), and
5. individuals with psoriasis and periodontitis (Psoriasis Periodontitis, PP). Levels of TNF-α, IL-17A, and YKL-40 will be measured in both saliva and serum samples. Additionally, correlations among these cytokines and between cytokine levels and clinical periodontal parameters-including Plaque Index (PI), Bleeding on Probing (BOP), Probing Pocket Depth (PPD), and Clinical Attachment Level (CAL)-will be analyzed.

Conclusion: The study is expected to provide insight into the immunological link between psoriasis and periodontal disease by evaluating TNF-α, IL-17A, and YKL-40 levels at both local (saliva) and systemic (serum) levels.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease affecting the supporting structures of the teeth, characterized by gingival inflammation, destruction of periodontal tissues, and alveolar bone loss. The disease primarily develops due to bacterial colonization at the tooth-gingival interface. Inflammatory mediators released in response to the interaction between a dysbiotic microbial biofilm and the host immune system play a critical role in tissue destruction and disease progression. Systemic conditions that affect the host immune system may exacerbate periodontal destruction in this multifactorial disease.

Psoriasis is a chronic inflammatory skin condition characterized by erythematous plaques or papules covered with silvery-white scales. The prevalence ranges between 1% and 3%, depending on the ethnic population, and it affects both genders equally. Although the exact etiopathogenesis of psoriasis remains unclear, several environmental and systemic factors-such as trauma, ultraviolet radiation, infections, medications, endocrine influences, psychological stress, alcohol consumption, and smoking-have been identified as potential triggers.

A possible association between psoriasis and periodontitis has been reported in multiple clinical studies and meta-analyses. Interleukin-17 (IL-17) is a pro-inflammatory cytokine that induces the expression of various inflammation-related mediators. It plays a central role in immune regulation and is implicated in inflammatory diseases, autoimmune disorders, and cancer. Elevated IL-17A levels have been detected in both psoriatic skin and serum samples of individuals with psoriasis when compared to healthy controls.

Tumor necrosis factor-alpha (TNF-α) is a polypeptide cytokine produced primarily by macrophages and monocytes. It functions as a multipotent regulator in immune responses by stimulating fibroblasts to release collagenase, increasing vascular permeability, promoting the release of other cytokines (such as IL-1α, IL-1β, IL-6, and IL-8), and enhancing the production of matrix metalloproteinases and adhesion molecules. TNF-α also synergizes with IL-1 to promote bone resorption. Elevated TNF-α levels in both serum and psoriatic lesions have been shown to decrease following effective treatment.

YKL-40 is a 40-kDa glycoprotein composed of tyrosine (Y), lysine (K), and leucine (L) at its N-terminal. It is secreted by neutrophils, macrophages, chondrocytes, synovial cells, osteoblasts, endothelial cells, and cancer cells. YKL-40 is associated with immune responses involving inflammation, tissue remodeling, and angiogenesis, and is considered an acute-phase protein.

A limited number of studies addressing the pathogenesis-related association between psoriasis and periodontal status have been identified in the literature, indicating a need for further investigation. To address this gap, a study is planned in which biomarkers associated with both periodontitis and psoriasis will be evaluated at both local and systemic levels.

The primary objective will be to comparatively assess TNF-α, IL-17A, and YKL-40 levels in saliva and serum samples of individuals with psoriasis, along with relevant clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria

* Voluntary participation
* No use of antibiotics within the past 6 months
* No periodontal treatment within the past 6 months
* Absence of systemic diseases known to affect periodontal health (e.g., diabetes, cardiovascular diseases)
* No infectious diseases such as tuberculosis, hepatitis, or AIDS
* Age 18 years or older
* Not pregnant (for female participants)

Exclusion Criteria:

* Pregnancy or ongoing lactation
* History of gingival treatment within the past 6 months
* History of any disease involving the oral mucosa (e.g., lichen planus, pemphigus vulgaris, chronic ulcerative stomatitis)
* Current use of systemic corticosteroids, immunosuppressive agents, or biological drugs
* History of systemic inflammatory diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, irritable bowel syndrome, diabetes mellitus)
* Fewer than 20 natural teeth (excluding third molars)
* Current smokers
* Age younger than 18 or older than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 participants are included after providing informed consent and meeting inclusion criteria. Participants are divided into five equal groups (n=20 per group):
  1. Systemically and periodontally healthy individuals (H),
  2. Systemically healthy individuals with gingivitis (Control Gingivitis, CG),
  3. Systemically healthy individuals with periodontitis (Control Periodontitis, CP),
  4. Individuals with psoriasis and gingivitis (Psoriasis Gingivitis, PG), and
  5. Individuals with psoriasis and periodontitis (Psoriasis Periodontitis, PP).
  Periodontal diagnoses are made based on the 2017 classification system of the American Academy of Periodontology (AAP) and the European Federation of Periodontology (EFP).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
TNF-α levels in saliva | at baseline (single visit)
  The level of tumor necrosis factor-alpha (TNF-α) in saliva, measured in picograms per milliliter (pg/mL), will be recorded at the initial visit.
TNF-α levels in serum | at baseline (single visit)
  The level of tumor necrosis factor-alpha (TNF-α) in serum, measured in picograms per milliliter (pg/mL), will be recorded at the initial visit.
IL-17A levels in saliva | at baseline (single visit)
  The level of interleukin-17A (IL-17A) in saliva, measured in picograms per milliliter (pg/mL), will be recorded at the initial visit.
IL-17A levels in serum | at baseline (single visit)
  The level of interleukin-17A (IL-17A) in serum, measured in picograms per milliliter (pg/mL), will be recorded at the initial visit
YKL-40 levels in saliva | at baseline (single visit)
  The level of YKL-40 in saliva, measured in picograms per milliliter (pg/mL), will be recorded at the initial visit.
YKL-40 levels in serum | at baseline (single visit)
  The level of YKL-40 in serum, measured in nanograms per milliliter (ng/mL), will be recorded at the initial visit.

SECONDARY OUTCOMES:
periodontal assesment | at baseline (single visit)
  probing pocket depth(PPD): Average probing pocket depth measured in millimeters at the initial visit.
Periodontal Assesment | Baseline (at single visit)
  Bleeding on Probing (BOP): Percentage of sites with bleeding on probing measured at the initial visit
Periodontal Assesment | Baseline (at single visit)
  Plaque Index (PI): Plaque Index score measured at the initial visit
Periodontal Assessment | Baseline (at single visit)
  Clinical Attachment Level (CAL): Clinical Attachment Level measured in millimeters at the initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Hazal DURMUS, DDS, Principal Investigator — Akdeniz Universty, Faculty Of Dentistry, Department Of Periodontology
Locations (1):
- Akdeniz University, Fculty of Dentistry, Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. Future data-sharing plans will depend on institutional policies, ethical considerations, and applicable regulatory requirements.

REFERENCES:
- [Background] Kong Y, Zhang S, Su X, Peng D, Su Y. Serum levels of YKL-40 are increased in patients with psoriasis: a meta-analysis. Postgrad Med. 2019 Aug;131(6):405-412. doi: 10.1080/00325481.2019.1643634. Epub 2019 Jul 22. PMID 31298974
- [Background] Martinez-Garcia M, Hernandez-Lemus E. Periodontal Inflammation and Systemic Diseases: An Overview. Front Physiol. 2021 Oct 27;12:709438. doi: 10.3389/fphys.2021.709438. eCollection 2021. PMID 34776994
- [Background] de Oliveira PS, Cardoso PR, Lima EV, Pereira MC, Duarte AL, Pitta Ida R, Rego MJ, Pitta MG. IL-17A, IL-22, IL-6, and IL-21 Serum Levels in Plaque-Type Psoriasis in Brazilian Patients. Mediators Inflamm. 2015;2015:819149. doi: 10.1155/2015/819149. Epub 2015 Aug 13. PMID 26351408
- [Background] Jimenez C, Carvajal D, Hernandez M, Valenzuela F, Astorga J, Fernandez A. Levels of the interleukins 17A, 22, and 23 and the S100 protein family in the gingival crevicular fluid of psoriatic patients with or without periodontitis. An Bras Dermatol. 2021 Mar-Apr;96(2):163-170. doi: 10.1016/j.abd.2020.08.008. Epub 2021 Jan 25. PMID 33531183
- [Background] Marruganti C, Gaeta C, Falciani C, Cinotti E, Rubegni P, Alovisi M, Scotti N, Baldi A, Bellan C, Defraia C, Fiorino F, Valensin S, Bellini E, De Rosa A, D'Aiuto F, Grandini S. Are periodontitis and psoriasis associated? A pre-clinical murine model. J Clin Periodontol. 2024 Aug;51(8):1044-1053. doi: 10.1111/jcpe.13996. Epub 2024 May 3. PMID 38699834